CLINICAL TRIAL: NCT00491751
Title: Clinical Utility of Endothelial Dysfunction in PAD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: H-23184
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2017-05

CONDITIONS: Peripheral Arterial Disease
Keywords: endothelium; nitric oxide; statins; ascorbic acid
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Atorvastatin; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Atorvastatin (Experimental): Atorvastatin 40 or 80 mg/day
  Interventions: Drug: atorvastatin
- Ascorbic Acid (Experimental): Ascorbic Acid 500 mg/day
  Interventions: Drug: ascorbic acid
- Placebo (Placebo Comparator): Placebo atorvastatin and Placebo ascorbic acid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: atorvastatin — atorvastatin 40 or 80 mg/day
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: ascorbic acid — ascorbic acid 500 mg/day
  Other Names: Vitamin C
  Arms: Ascorbic Acid
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
This study will seek to determine whether non-invasive measures of endothelial function have utility as surrogate markers of cardiovascular risk in patients with peripheral arterial disease undergoing vascular surgery. Measurements of endothelial function will be made before and after initiation of atorvastatin, ascorbic acid, or placebo therapy during the pre-operative period. We will then examine cardiovascular events following surgery. We hypothesize that patients who have no improvement in endothelial function will have increased cardiovascular risk compared to patients with improvement in endothelial function.

DETAILED DESCRIPTION:
Part 1 of the study will involve only patients with PAD who are undergoing non-cardiac surgery and is an intervention study. Part 2 will involve patients with PAD who have participated in Part 1 and patients with PAD who are not undergoing surgery. This part of the study does not involve an intervention.

The protocol for patients undergoing surgery is as follows: Part 1. Intervention study with follow-up for 30 days after surgery. Patients with planned surgery will be enrolled. We will test endothelial function at baseline using ultrasound and tonometry. They will then be randomzied to one of three groups: Atorvastatin 80 mg/d, Vitamin C 500 mg/d, or placebo. Subjects already on a statin medication at the time of enrollment will receive 40 mg/d of atorvastatin. Patients taking high dose statin (>40 mg/day) will be randomized to received vitamin C or placebo, and will not be eligible to receive any additional statin as part of the study. In the week immediately prior to surgery, we will test endothelial function a second time. They will then be followed for 30 days beginning with the day of surgery for cardiovascular events. Part 1 of the study involves 4 visits as follows: Visit 1 at enrollment will take place within 7-30 days of non-emergent vascular surgery and will last approximately 60 minutes Visit 2 will take place within approximately 1 week of surgery and will last approximately 30-40 minutes Visit 3 will occur on the 1st post-operative day and will last approximately 10-15 minutes Visit 4 will take place only if the subject is still an in-patient. It will take approximately 10-15 minutes Telephone contact will occur at 30 days post surgery and every six months thereafter for two years. The duration of telephone follow-up is expected to be approximately 5-10 minutes. Part 2 (long term follow-up): Patients who have completed Part 1 will be continued on in Part 2 of the study. Part 2 involves two year follow-up with no study medication. Telephone contact will be made every 6 months. subjects will make a visit to our research unit one year after the initial visit for physical examination, and if applicable, an ultrasound study of their bypass grafts.

The protocol for patients with PAD who are not undergoing surgery is as follows. These patients will participate in Part 2 of the study only (long-term follow-up with no intervention). Visit 1: will last approximately 60 minutes and involve measurement of endothelial function by ultrasound and tonometry. We will contact the subject every 6 months by telephone (5-10 minutes) for two years to determine whether a cardiovascular event has occurred. Visit 2 will occur at 1 year post enrollment and will last approximately 20-30 minutes. If the subject has had peripheral bypass surgery, we will perform an ultrasound study to determine graft blood flow.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 21-99 years old.
2. Peripheral Arterial Disease. PAD is defined clinically and by angiography, magnetic resonance imaging, vascular ultrasound, or ankle brachial index less than 0.9.
3. Able to provide informed consent and complete the study procedure.
4. Patients undergoing non-emergent vascular surgery (peripheral arterial bypass, abdominal aortic aneurysm repair, carotid endarterectomy, or limb amputation) or other non-cardiac surgery.

Exclusion Criteria:

1. Emergent or urgent surgery that must be performed sooner than one week after enrollment
2. Unstable angina, myocardial infarction, stroke, coronary revascularization, or decompensated heart failure within 1 month of enrollment. Patients who require cardiac catheterization and surgical or percutaneous coronary revascularization prior to vascular surgery will be excluded.
3. Clinically evident major illness of other organ systems, including cancer, end-stage renal disease, hepatic failure, or other conditions that make participation inappropriate.
4. Women who are lactating, pregnant, or of childbearing potential and not using a reliable contraceptive method. Pregnancy will be excluded by a urine pregnancy test.
5. Patients with liver function tests or serum creatine kinase >3 times the upper limit of normal.
6. Patients who have received an investigational drug within 30 days of enrollment.
7. Patients or subjects with a history of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
8. Known occlusive atherosclerosis of the subclavian artery or upper extremity, because such disease will interfere with induction of reactive hyperemia during the brachial artery ultrasound studies.
9. Patients will be excluded if they are taking vitamin C in a dose greater than 2 times the Recommended Daily Allowance (>120 mg/day) within 1 month of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2004-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Hamburg, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: May 2004 to June 2010.
Groups:
- Atorvastatin: Atorvastatin 40 or 80 mg
- Ascorbic Acid: Ascorbic Acid 500 mg per day
Period: Overall Study
Arm/Group | Atorvastatin | Ascorbic Acid | Placebo
Started | 22 | 44 | 42
Completed | 22 | 44 | 42
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Ascorbic Acid | Placebo | Total
Number analyzed (Participants) | 22 | 44 | 42 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 22 | 21 | 54
  >=65 years | 11 | 22 | 21 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (11) | 66 (8) | 65 (9) | 66 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 6 | 29
  Male | 13 | 30 | 36 | 79
Region of Enrollment [Number; unit: participants]
  United States | 22 | 44 | 42 | 108

OUTCOME MEASURES:

1. Primary Outcome: Change in FMD
Description: Change in flow mediated dilation with treatment: FMD visit 2 - FMD visit 1 FMD is measured by using vascular ultrasound to determine the baseline diameter of the brachial artery. Endothelium-dependent vasodilation is induced by 5-minute arterial occlusion with a blood pressure cuff. When the cuff is released, the resultant increase in blood flow (reactive hyperemia) stimulates vasodilation of the brachial artery. This flow-mediated dilation (FMD) is expressed as the percent change from baseline. Healthy individuals typical dysplay a 10 to 12% dilation. Individuals with PAD had markedly impaired dilation of 6-7. The currernt study sought to determine whether a change in FMD would occur following intervention.
Time Frame: 1-4 weeks
Population: All enrolled subjects were analyzed.
Measure: Mean (Standard Deviation); unit: percent change of FMD
Arm/Group | Atorvastatin | Ascorbic Acid | Placebo
Number analyzed (Participants) | 22 | 44 | 42
percent change of FMD | 0.88 (3.0) | 0.41 (3.6) | 0.88 (3.5)

2. Secondary Outcome: Percentage Change in FMD in All Participants With and Without a CVD Event (Not by Treatment Group)
Description: This outcome is independent of the treatment group so the groups are 'CVD event' and ' No CVD Event'. Cardiovascular events (CVD) included cardiovascular disease, myocardial infarction, congestive heart failure, stroke, and unstable angina.
Time Frame: 2 months
Population: For this outcome all participants were stratified into 2 groups: those with, and those without a CVD event (not by treatment group)
Measure: Mean (Standard Deviation); unit: percent change of flow-mediated dilation
Groups:
- CVD Event: All subjects with a cardiovascular event regardless of treatment group.
- No CVD Event: All subjects without a cardiovascular event regardless of treatment group.
Arm/Group | CVD Event | No CVD Event
Number analyzed (Participants) | 16 | 92
percent change of flow-mediated dilation | 0.5 (4.0) | 0.7 (3.4)

ADVERSE EVENTS:
Time Frame: 2 months
Description: All subjects were followed for 2 months. They were questioned about adverse events and medical records were reviewed.
Groups:
- Ascorbic Acid: Ascorbi acid 500 mg [per day
- Placebo: Placebo for atorvastatin and ascorbic acid
Arm/Group | Atorvastatin | Ascorbic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 1/44 | 1/42
Serious Adverse Events (participants affected / at risk) | 3/22 | 6/44 | 7/42
Other Adverse Events (participants affected / at risk) | 0/22 | 0/44 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=22) | Ascorbic Acid (N=44) | Placebo (N=42)
Myocardial infaction (Cardiac disorders) | 2 | 2 | 6
Unstable angina (Cardiac disorders) | 0 | 0 | 3
Congestive heart failure (Cardiac disorders) | 0 | 2 | 2
CVA/TIA (Nervous system disorders) | 2 | 2 | 0
Venticular fibrillation (Cardiac disorders) | 0 | 0 | 1
Other CVD event (Cardiac disorders) | 1 | 3 | 3

LIMITATIONS AND CAVEATS:
The study was terminated after enrollment of 108 of 450 subjects due to inability to enroll a sufficient number of subjects. Enrollment was difficult because nearly all potential subjects were already taking a statin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No